CLINICAL TRIAL: NCT04642001
Title: Association of Two Desensitizing Protocols to Control Dentinal Hypersensitivity in Non-carious Lesions: A Randomized, Double-blind Clinical Trial.
Brief Title: Association of Two Desensitizing Protocols to Control Dentinal Hypersensitivity in Non-carious Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Para (Other)
Responsible Party: Principal Investigator, Cecy Martins Silva, clinical professor, Universidade Federal do Para
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: UFPara-009
Record Dates: First submitted 2020-11-11; First posted 2020-11-24 (Actual); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: Dental Hypersensitivity
MeSH Terms: interventions — halofantrine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group G1 (Other): Photon Laser III-DMC (without radiation emission) + My First- Colgate
  Interventions: Other: Photon Laser III-DMC (without radiation emission) + My First- Colgate
- Group G2 (Experimental): Photon Laser III-DMC (without radiation emission) + Sensodyne® Rápido Alívio/GSK
  Interventions: Other: Photon Laser III-DMC (without radiation emission) + Sensodyne® Rapid Relief / GSK
- Group G3 (Experimental): Photon Laser III-DMC (with irradiation emission) + My First- Colgate
  Interventions: Radiation: Photon Laser III-DMC (with irradiation emission) + My First- Colgate
- Group G4 (Experimental): Photon Laser III-DMC (with irradiation emission) + Sensodyne® Rápido Alívio/GSK
  Interventions: Combination Product: Photon Laser III-DMC (with irradiation emission) +Sensodyne® Rapid Relief / GSK

INTERVENTIONS:
Other: Photon Laser III-DMC (without radiation emission) + My First- Colgate — Positioning of the FBM (Photon Laser III / DMC) without emitting radiation, the equipment's sound was mimicked with the Beep application (Foncannon Inc, Google, © 2018), followed by the use of fluoride-free toothpaste (My First- Colgate) and brushing three times a day.
  Arms: Group G1
Other: Photon Laser III-DMC (without radiation emission) + Sensodyne® Rapid Relief / GSK — Positioning of FBM (Photon Laser III / DMC) without emitting radiation, the equipment's sound was mimicked with the Beep application (Foncannon Inc, Google, © 2018), followed by the application of toothpaste containing strontium acetate (Sensodyne® Rapid Relief / GSK) and brushing three times a day.
  Arms: Group G2
Radiation: Photon Laser III-DMC (with irradiation emission) + My First- Colgate — Emission of FBM therapy (Photon Laser III / DMC), followed by the use of fluoride-free toothpaste (My First- Colgate) and brushing three times a day.
  Arms: Group G3
Combination Product: Photon Laser III-DMC (with irradiation emission) +Sensodyne® Rapid Relief / GSK — Emission of FBM therapy (Photon Laser III / DMC), followed by the application of toothpaste containing strontium acetate (Sensodyne® Rapid Relief / GSK) and brushing three times a day.
  Arms: Group G4

SUMMARY:
This randomized, double-blind clinical trial evaluated the effect of photobimodulation associated with 8% strontium acetate in the treatment of dentin hypersensitivity in non-carious lesions and analyzed the risk factors with the patient's quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 to 50 years
* Good general health
* Dental sensitivity with response ≥ 4 on the 10 cm long visual analog scale (EVA)
* Presence of at least two hypersensitive teeth with a depth of up to 1 mm (measured with a millimeter probe)
* Exposed root surface caused by abrasion, erosion or gum recession

Exclusion Criteria:

* Volunteers using analgesic medication
* Presence of teeth with evidence of carious lesions, pulpitis, defective restorations and moderate or severe periodontal disease
* Patients who had undergone any whitening therapy or professional or homemade desensitizer in the last six months
* Patient with fixed orthodontic appliances
* Drug users or pregnant women were also excluded.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2019-08-07 (Actual); Primary Completion 2020-09-15 (Actual); Study Completion 2020-11-05 (Actual)

PRIMARY OUTCOMES:
dentin sensitivity | 30 days after the end of treatment
  evaluation of dentinal sensitivity during treatment and one month after its end, by means of tactile and evaporative stimuli according to the visual analog scale with values from 0 to 10, with higher values indicating a worse level of pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Federal do Pará, Belém, Pará, Brazil